CLINICAL TRIAL: NCT01444378
Title: Absolute Pro® Peripheral Self-Expanding Stent System and the Absolute Pro® LL Peripheral Self-Expanding Stent Systems in the Treatment of Subjects With Atherosclerotic De Novo or Restenotic Lesions in the Native Superficial Femoral Artery and/or Native Proximal Popliteal Artery.
Brief Title: Absolute Pro® MOMENTUM™
Acronym: MOMENTUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-110
Record Dates: First submitted 2011-09-21; First posted 2011-09-30 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease
Keywords: Atherosclerosis; Claudication; Peripheral Arterial Occlusive Disease; Stent
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Atherosclerosis; Intermittent Claudication; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Absolute Pro® and Pro LL® Peripheral Stent Systems (Experimental)
  Interventions: Device: Stenting using Absolute Pro® and Pro LL® Peripheral Stent Systems

INTERVENTIONS:
Device: Stenting using Absolute Pro® and Pro LL® Peripheral Stent Systems — Stenting of the Superficial Femoral Artery (SFA) and/or proximal popliteal artery using either of these devices.

SUMMARY:
To evaluate the safety and effectiveness of the Absolute Pro® Peripheral Self-Expanding Stent System and the Absolute Pro® LL Peripheral Self-Expanding Stent System for the treatment of subjects with atherosclerotic de novo or restenotic lesions in the native superficial femoral artery (SFA) and/or the native proximal popliteal artery (PPA).

CAUTION: Absolute Pro® Peripheral Self-Expanding Stent System and the Absolute Pro® LL Peripheral Self-Expanding Stent Systems are investigational devices. Limited by Federal (U.S.) law to investigational use only.

ELIGIBILITY:
General Clinical Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and is able to provide informed consent.
3. Subject agrees to undergo all protocol-required follow-up examinations and requirements at the investigational site.
4. Subject is diagnosed as having moderate to severe claudication (Rutherford-Becker Clinical Category 2-3) or ischemic rest pain (Rutherford-Becker Clinical Category 4).
5. Female subject of childbearing potential must:

   * have had a negative pregnancy test (serum HCG) within 14 days before treatment;
   * not be nursing at the time of treatment; and
   * agree at time of consent to use birth control during participation in this trial.
6. Subject has life expectancy > 12 months.

Angiographic Inclusion Criteria:

1. A single de novo or restenotic [not previously treated with stent, brachytherapy, laser, surgical bypass, or endarterectomy] native disease segment of the superficial femoral artery (SFA) and/or proximal popliteal artery (PPA) located within the following parameters: ≥1 cm below the femoral bifurcation in the SFA. ≥3 cm above the proximal margin of the intercondylar fossa.
2. Disease segment length visually estimated to be ≤ 14 cm (140 mm) and can be treated with one stent.
3. Disease segment visually estimated to be ≥ 50% stenosis or a total occlusion.
4. Target vessel reference diameter visually estimated to be ≥ 4.0 mm and ≤ 7.0 mm.
5. A patent ipsilateral iliac artery, defined as < 50% stenosis, as confirmed by arteriography.
6. At least one patent distal outflow artery (anterior tibial, posterior tibial, peroneal) defined as < 50% stenosis, that provides in-line circulation to the lower leg and foot.
7. Total occlusion length ≤ 8 cm.

General Clinical Exclusion Criteria:

1. Subject is unable to walk.
2. Subject has undergone any non-iliac percutaneous intervention, e.g. coronary, carotid, < 30 days prior to the planned index procedure.
3. Subject has received, or is on the waiting list for, a major organ transplant.
4. Subject is diagnosed as Rutherford-Becker Clinical Category 5 or 6 in either extremity.
5. Subject is diagnosed as Rutherford-Becker Clinical Category 0 or 1 in the target extremity (i.e., where the investigational stent will be placed).
6. Subject has elevated serum creatinine > 2.5 mg/dl.
7. Subject is on chronic hemodialysis.
8. Subject has documented or suspected uncontrolled diabetes mellitus (DM), unless HbA1c has been assessed as < 7.0% within 3 months prior to index procedure.
9. Subject has had a myocardial infarction (MI) within the previous 30 days of the planned index procedure.
10. Subject has had a stroke within the previous 30 days of the planned index procedure and/or has deficits from a prior stroke that limits the subject's ability to walk.
11. Subject has unstable angina defined as rest angina with ECG changes.
12. Subject has a groin infection, or an acute systemic infection that has not been treated successfully or is currently under treatment.
13. Subject has acute thrombophlebitis or deep vein thrombosis in either extremity.
14. Subject is unable to take required antiplatelet therapy or requires any planned procedure that would necessitate the discontinuation of clopidogrel, prasugrel, ticagrelor or ticlopidine within 30 days following the procedure.
15. Subject has other medical illnesses (e.g., cancer or congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation or is associated with limited life-expectancy, i.e., less than 1 year.
16. Subject is currently participating in an investigational drug, biologic, or device study.
17. Subject is unable to understand or unwilling to cooperate with study procedures.
18. Subject is allergic to nickel, titanium, platinum, contrast media, or any study-required medication that is not amenable to pre-treatment.
19. Subject has a known bleeding or hypercoagulability disorder or significant anemia (Hgb < 8.0) that cannot be corrected.
20. Subject requires general anesthesia for the procedure.
21. Subject has ischemic or neuropathic ulcers on either foot.
22. Subject has had any type of amputation to the ipsilateral extremity, or a contralateral extremity amputation other than of the toe or forefoot.
23. Subject is part of a vulnerable population who, in the judgment of the investigator, is unable to give informed consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention.

Angiographic Exclusion Criteria:

1. Total occlusion of the ipsilateral iliac artery.
2. Target extremity has multilevel disease that requires other staged procedures within 30 days before or after the procedure.
3. Target extremity has been previously treated with any of the following: surgical bypass or endarterectomy.
4. Target vessel has an angiographically significant (> 50% DS) lesion located distal to the target lesion that requires treatment at the time of the index procedure or by a staged procedure within 30 days before or after the procedure.
5. Target vessel has been previously treated at any location with a stent, or has been previously treated ≤ 5 cm from the proximal or distal margin of the target lesion with brachytherapy or laser.
6. Target lesion is within or adjacent to an aneurysm.
7. Target lesion or vessel has angiographic evidence of thrombus that is unresponsive to anti-thrombotic therapies.
8. Subject has a contralateral superficial femoral or proximal popliteal artery lesion that requires treatment within 30 days before or after the procedure.
9. Subject has a history of aortic revascularization or has an abdominal aortic aneurysm > 3 cm.
10. Subject has evidence of thromboembolism or atheroembolism from treatment of an ipsilateral iliac lesion.
11. .Subject has any condition that precludes safe access to the target lesion or target vessel, e.g. severe calcification, excessive tortuosity.
12. Target lesion requires use of re-entry, ablative, cutting balloon, atherectomy, or similar devices to cross or treat the lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce H. Gray, DO, Principal Investigator — University Medical Center Greenville
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was registered in the MOMENTUM trial on November 2011. Enrollment in the trial was closed on November 2013. Based on the February 19, 2015, data extraction, 141 patients were registered in the MOMENTUM trial.at 32 US sites
Period: Overall Study
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Started | 141 (A total of 141 patients were enrolled into MOMENTUM)
Completed | 124
Not Completed | 17
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3
Not completed — Administrative Closure Of The Study | 2
Not completed — Missed Visits | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 88
Race/Ethnicity, Customized [Number; unit: participants] — Subjects who are in multiple race categories are counted in each checked category. The sum of the percentages of all race categories may not equal 100%.
  participants
    American Indian or Alaska Native | 0
    Asian | 1
    Black or African Heritage | 19
    Latino-Hispanic | 3
    Native Hawaiian or Other Pacific Islander | 0
    White | 120
Region of Enrollment [Number; unit: participants]
  United States | 141

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event (MAE)
Description: Primary safety endpoint is freedom from MAE which is defined as a composite of:
  * Death due to all causes
  * Index limb major amputation (at or above the ankle)
  * Clinically-driven target lesion revascularization (TLR)
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants
  Death due to all causes | 0.0
  Index Limb Major Amputation (at or above the ankle | 0.0
  Clinically-driven TLR | 0.0

2. Primary Outcome: Freedom From Vessel Patency
Description: This is the primary effectiveness endpoint which is defined as the absence of in-stent restenosis (≥ 50%) as determined by duplex ultrasonography or arteriography and without clinically driven TLR. The vessel patency rate was estimated by the Kaplan-Meier method with the standard error estimated using the Greenwood formula.
Time Frame: 0 to 365 days
Population: Intention-to-treat (ITT) population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 60.8

3. Secondary Outcome: Acute Success : Device Success
Description: Device success defined on a per device basis, as the achievement of successful delivery and deployment of the trial device at the intended target lesion and successful withdrawal of the delivery catheter.
Time Frame: With in 2 days of index post procedure
Population: ITT population, per device analysis.
Measure: Number; unit: percentage of devices
Units Other Than Participants: Device
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
Number analyzed (Device) | 146
percentage of devices | 96.6

4. Secondary Outcome: Acute Success : Clinical Success
Description: Clinical success: Defined on a per patient basis, as the attainment of a final residual stenosis of < 30% by core laboratory assessment using the study device(s) and/or any adjunctive device at all intended target lesion(s) without complications within 2 days after the index procedure or at hospital discharge, whichever is sooner.
Time Frame: With in 2 days after index post procedure or at hospital discharge (before 1 month)
Population: ITT population, per subject analysis
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 137
percentage of participants | 97.1

5. Secondary Outcome: Acute Success : Technical Success
Description: Technical success: Device success plus attainment of final residual stenosis of < 30%
Time Frame: With in 2 days of index post procedure
Population: ITT population, per lesion analysis
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Target Lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 137
Number analyzed (Target Lesions) | 137
percentage of target lesions | 97.1

6. Secondary Outcome: Freedom From Vessel Patency
Description: as for outcome 2
Time Frame: 0 to 30 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

7. Secondary Outcome: Freedom From Vessel Patency
Description: as for outcome 2
Time Frame: 0 to 180 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 90.0

8. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: A measure of the fall in blood pressure in the arteries supplying the legs and is used to detect evidence of blockages in the peripheral vessels. It is calculated by dividing the higher systolic blood pressure in the ankle (dorsalis pedis or posterior tibial) of the one leg by the higher of the two systolic blood pressures in the arms.
  ABI=Highest Ankle Systolic Pressure/Highest Brachial Systolic Pressure. The ABI is the ratio of the ankle to arm pressure, and an ABI between 0.9 and 1.3 is considered normal. A reduced ABI (less than 0.9) is consistent with peripheral artery occlusive disease, with values below 0.8 indicating moderate disease and below 0.5 severe disease.
  A value greater than 1.3 is considered abnormal suggesting calcification of the walls of the arteries and noncompressible vessels, reflecting severe peripheral vascular disease. For patients in whom the ABI cannot be accurately measured , toe pressure measurement and toe brachial index should be used.
Time Frame: Pre-Procedure
Population: ITT population, per subject analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point. ABI > 1.3 was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 136
Ratio | 0.75 (0.19)

9. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 8
Time Frame: 1 month
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 110
Ratio | 0.97 (0.13)

10. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 118
Ratio | 0.92 (0.18)

11. Secondary Outcome: Ankle Brachial Index (ABI) for the Treated Limb
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 106
Ratio | 0.88 (0.17)

12. Secondary Outcome: Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Revascularization within the borders of the stent, +5 mm unstented vessel at both ends, with diameter stenosis ≥ 50% (determined by duplex ultrasound or angiographic core laboratory) (Note: This does not include coincidental overlap of a percutaneous transluminal angioplasty (PTA) balloon or stent into a study stent, that has <50% stenosis, while treating a non-target lesion in the target vessel) plus one or both of the following:
  * Worsening Rutherford-Becker Clinical Category;
  * Change in ABI by >0.15 and ABI ≤0.8
Time Frame: At 1 month
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

13. Secondary Outcome: Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 12
Time Frame: At 6 months
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 7.1

14. Secondary Outcome: Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 12
Time Frame: At 1 year
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 19.1

15. Secondary Outcome: Any Target Lesion Revascularization (TLR)
Description: TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be prospectively classified as clinically-driven or not clinically-driven by the investigator prior to repeat angiography. An independent angiographic core laboratory will verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Time Frame: At 1 month
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

16. Secondary Outcome: Any Target Lesion Revascularization (TLR)
Description: as for outcome 15
Time Frame: At 6 months
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 1.4

17. Secondary Outcome: Any Target Lesion Revascularization (TLR)
Description: as for outcome 15
Time Frame: At 1 year
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 3.5

18. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the ipsilateral superficial femoral artery and the proximal popliteal artery, including the target lesion itself.
Time Frame: At 1 month
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

19. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 18
Time Frame: At 6 months
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 5.0

20. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 18
Time Frame: At 1 year
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 7.8

21. Secondary Outcome: Death
Time Frame: At 1 month
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

22. Secondary Outcome: Death
Time Frame: At 6 months
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.7

23. Secondary Outcome: Death
Time Frame: At 1 year
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 2.1

24. Secondary Outcome: Freedom From Stent Patency
Description: Primary Stent Patency defined as < 50% stenosis of the stented segment, as determined by duplex ultrasound or arteriography.
Time Frame: 0 to 30 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

25. Secondary Outcome: Freedom From Stent Patency
Description: as for outcome 24
Time Frame: 0 to 180 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 90.0

26. Secondary Outcome: Freedom From Stent Patency
Description: as for outcome 24
Time Frame: 0 to 365 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 60.8

27. Secondary Outcome: Freedom From Stent Patency
Description: as for outcome 24
Time Frame: 0 to 379 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 53.0

28. Secondary Outcome: Freedom From Any Ipsilateral Amputation
Description: Amputation is defined as the removal of a body extremity by surgery. For this trial, the definition of amputation will only include amputations of the limb that was treated. A minor amputation will be defined as below the ankle; a major amputation will be defined as at or above the ankle.
Time Frame: At day 0 (on the day of index procedure)
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

29. Secondary Outcome: Freedom From Any Ipsilateral Amputation
Description: as for outcome 28
Time Frame: 0 to 30 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

30. Secondary Outcome: Freedom From Any Ipsilateral Amputation
Description: as for outcome 28
Time Frame: 0 to 180 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

31. Secondary Outcome: Freedom From Any Ipsilateral Amputation
Description: as for outcome 28
Time Frame: 0 to 365 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

32. Secondary Outcome: Freedom From Any Ipsilateral Amputation
Description: as for outcome 28
Time Frame: 0 to 379 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

33. Secondary Outcome: Embolic Events in the Treated Limb (as Reported by Site)
Description: Embolic Event is defined as formation of a thrombus within the target lesion or stent with migration or atherosclerotic emboli migration to a distal artery.
Time Frame: At 1 month
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.7

34. Secondary Outcome: Embolic Events in the Treated Limb (as Reported by Site)
Description: as for outcome 33
Time Frame: At 6 months
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 1.4

35. Secondary Outcome: Embolic Events in the Treated Limb (as Reported by Site)
Description: as for outcome 33
Time Frame: At 1 year
Population: ITT population, per subject analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 1.4

36. Secondary Outcome: Rutherford-Becker Clinical Category for the Treated Limb
Description: The Rutherford Becker clinical category is a scale to measure chronic limb ischemia.
  Category and Clinical Description:
  0 = Asymptomatic, no hemodynamically significant occlusive disease, 1 = Mild claudication, 2 = Moderate claudication, 3 = Severe claudication, 4 = Ischemic rest pain, 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable.
Time Frame: Pre-procedure
Population: ITT population, per subject analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 136
percentage of participants
  Category 0 | 0.0
  Category 1 | 0.0
  Category 2 | 27.9
  Category 3 | 62.5
  Category 4 | 9.6
  Category 5 | 0.0
  Category 6 | 0.0

37. Secondary Outcome: Rutherford-Becker Clinical Category for the Treated Limb
Description: as for outcome 36
Time Frame: 1 month
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 116
percentage of participants
  Category 0 | 56.0
  Category 1 | 24.1
  Category 2 | 18.1
  Category 3 | 1.7
  Category 4 | 0.0
  Category 5 | 0.0
  Category 6 | 0.0

38. Secondary Outcome: Rutherford-Becker Clinical Category for the Treated Limb
Description: as for outcome 36
Time Frame: 6 months
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 116
percentage of participants
  Category 0 | 50.9
  Category 1 | 21.6
  Category 2 | 15.5
  Category 3 | 12.1
  Category 4 | 0.0
  Category 5 | 0.0
  Category 6 | 0.0

39. Secondary Outcome: Rutherford-Becker Clinical Category for the Treated Limb
Description: as for outcome 36
Time Frame: 12 months
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 104
percentage of participants
  Category 0 | 52.9
  Category 1 | 23.1
  Category 2 | 19.2
  Category 3 | 4.8
  Category 4 | 0.0
  Category 5 | 0.0
  Category 6 | 0.0

40. Secondary Outcome: Walking Impairment Questionnaire Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ), a disease-specific instrument utilized to characterize walking ability through a questionnaire as an alternative to treadmill testing. It is a measure of subject-perceived walking performance for subjects with Peripheral Artery Disease (PAD) and/or intermittent claudication. The WIQ quantifies patient-reported walking speed, walking distance, and stair-climbing ability, respectively, on a scale of 0 (= worst) to 100 (= best). The highest possible score for each domain is 100%, which indicates no difficulty. Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Time Frame: Pre-procedure
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Walking Distance Score; Walking Speed Score; Stair Climbing Score: Stenting using Absolute Pro® and Pro LL® Peripheral Stent Systems: Stenting of the Superficial Femoral Artery (SFA) and/or proximal popliteal artery using either of these devices.
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 140 | 140 | 138
scores on a scale | 15.94 (18.71) | 20.45 (20.31) | 28.20 (26.85)

41. Secondary Outcome: Walking Impairment Questionnaire Scores
Description: as for outcome 40
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 120 | 120 | 114
scores on a scale | 47.82 (36.74) | 46.19 (32.11) | 54.53 (35.20)

42. Secondary Outcome: Walking Impairment Questionnaire Scores
Description: as for outcome 40
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 124 | 124 | 123
scores on a scale | 49.61 (38.67) | 44.89 (31.82) | 55.05 (35.56)

43. Secondary Outcome: Walking Impairment Questionnaire Scores
Description: as for outcome 40
Time Frame: 12 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Walking Distance Score | Walking Speed Score | Stair Climbing Score
Number analyzed (Participants) | 111 | 110 | 111
scores on a scale | 48.32 (37.53) | 42.92 (32.35) | 52.59 (35.64)

44. Secondary Outcome: Maximum Walking Distance
Time Frame: Pre-procedure
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 140
percentage of participants
  0 feet | 0.0
  20 feet | 3.6
  50 feet | 12.9
  150 feet | 21.4
  300 feet | 13.6
  600 feet | 12.1
  900 feet | 12.1
  1500 feet | 24.3

45. Secondary Outcome: Maximum Walking Distance
Time Frame: 1 month
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 120
percentage of participants
  0 feet | 0.0
  20 feet | 1.7
  50 feet | 4.2
  150 feet | 4.2
  300 feet | 14.2
  600 feet | 10.0
  900 feet | 10.8
  1500 feet | 55.0

46. Secondary Outcome: Maximum Walking Distance
Time Frame: 6 months
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 124
percentage of participants
  0 feet | 0.8
  20 feet | 2.4
  50 feet | 6.5
  150 feet | 7.3
  300 feet | 8.1
  600 feet | 6.5
  900 feet | 7.3
  1500 feet | 61.3

47. Secondary Outcome: Maximum Walking Distance
Time Frame: 12 months
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
percentage of participants
  0 feet | 0.9
  20 feet | 0.9
  50 feet | 6.3
  150 feet | 6.3
  300 feet | 9.0
  600 feet | 8.1
  900 feet | 6.3
  1500 feet | 62.2

48. Secondary Outcome: Stent Integrity by X-ray
Description: Xrays were performed to evaluate stent integrity and to determine the presence of any stent fractures.
  Grade of fracture as follows:
  0 - No stent fracture(s) identified
  1. - Single strut fracture only
  2. - Multiple strut fractures
  3. - Stent fracture with alignment
  4. - Fracture out of alignment (≥ 2 segments)
  5. - Spiral Fracture
Time Frame: 12 months
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 106
percentage of participants
  0 - No Fracture | 95.3
  1 - Single Strut | 1.9
  2 - Multiple Struts | 2.8
  3 - Stent Fracture w/Alignment | 0.0
  4 - Stent Fracture out of Alignment (2+ segments) | 0.0
  5 - Spiral Fracture | 0.0

49. Secondary Outcome: Toe Brachial Index (TBI)
Description: The toe brachial index is the ratio of the resting ipsilateral toe systolic blood pressure as compared to the highest resting brachial systolic blood pressure. A normal range is 0.9 to 1.3.
Time Frame: At 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 23
ratio | 0.73 (0.19)

50. Secondary Outcome: Toe Brachial Index (TBI)
Description: as for outcome 49
Time Frame: At 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 18
ratio | 0.70 (0.24)

51. Secondary Outcome: Toe Brachial Index (TBI)
Description: as for outcome 49
Time Frame: At 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 21
ratio | 0.71 (0.22)

52. Secondary Outcome: Duplex Ultrasound: Maximum In-Stent Peak Systolic Velocity (PSV)
Description: In-Stent Restenosis:
  Re-narrowing within the margins of the stent following the reduction of a previous narrowing. It is defined as the presence of a hemodynamically significant restenosis (≥ 50%), as determined by duplex ultrasound or arteriography.
Time Frame: 1 month
Population: ITT population, per lesion analysis. In-stent peak systolic velocity (PSV) and in-stent peak systolic velocity ratio (PSVR) are excluded from the analysis, for subjects who had TLR prior to the duplex ultrasound or duplex ultrasound was out of the protocol defined window or duplex ultrasound was not readable.
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 114
Number analyzed (Target lesions) | 114
cm/sec | 142.8 (40.4)

53. Secondary Outcome: Duplex Ultrasound: Maximum In-Stent Peak Systolic Velocity (PSV)
Description: as for outcome 52
Time Frame: 12 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 87
Number analyzed (Target lesions) | 87
cm/sec | 214.7 (105.0)

54. Secondary Outcome: Duplex Ultrasound: In-Stent Peak Systolic Velocity Ratio (PSVR)
Description: In-Stent Restenosis: Re-narrowing within the margins of the stent following the reduction of a previous narrowing. It is defined as the presence of a hemodynamically significant restenosis (≥ 50%), as determined by duplex ultrasound or arteriography. A PSVR of > 2.4 will be used to determine restenosis via duplex ultrasound.
Time Frame: 1 month
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 113
Number analyzed (Target lesions) | 113
cm/sec | 1.13 (0.28)

55. Secondary Outcome: Duplex Ultrasound: In-Stent Peak Systolic Velocity Ratio (PSVR)
Description: as for outcome 54
Time Frame: 12 months
Population: as for outcome 52
Measure: Mean (Standard Deviation); unit: cm/sec
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 85
Number analyzed (Target lesions) | 85
cm/sec | 1.98 (1.24)

56. Secondary Outcome: Acute Stent Thrombosis
Description: Stent thrombosis was defined as total occlusion identified within the stent by arteriography and/or ultrasound that occurs within 30 days post-index procedure.
Time Frame: 0 - 24 Hours Post Study Procedure
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

57. Secondary Outcome: Sub-Acute Stent Thrombosis
Description: as for outcome 56
Time Frame: > 24 Hours - 30 Days Post Study Procedure
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 0.0

58. Secondary Outcome: Stent Occlusion
Description: Stent occlusion was defined as total occlusion identified within the stent by arteriography and/or ultrasound that occurs > 30 days post-index procedure.
Time Frame: > 30 Days Post Study Procedure
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 10.6

59. Secondary Outcome: In-Segment Percent Diameter Stenosis (%DS)
Description: Percent Diameter Stenosis:
  The value calculated as 100 * (1 - Minimum Lumen Diameter/Reference Vessel Diameter) using the mean values from two orthogonal views (when possible) by Quantitative Analysis.
Time Frame: Pre-Procedure
Population: ITT population, per lesion analysis. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 137
Number analyzed (Target lesions) | 137
Percent Diameter stenosis | 79.02 (16.90)

60. Secondary Outcome: In-Segment Percent Diameter Stenosis (%DS)
Description: as for outcome 59
Time Frame: Post-Procedure (≥ 1 day)
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 137
Number analyzed (Target lesions) | 137
Percent Diameter stenosis | 15.18 (8.91)

61. Secondary Outcome: In-Stent Percent Diameter Stenosis (%DS)
Description: as for outcome 59
Time Frame: Post-Procedure (≥ 1 day)
Population: as for outcome 59
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 137
Percent Diameter stenosis | 4.10 (13.05)

62. Secondary Outcome: Freedom From Ipsilateral Major Amputation
Description: as for outcome 28
Time Frame: At day 0 (on the day of index procedure)
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

63. Secondary Outcome: Freedom From Ipsilateral Major Amputation
Description: as for outcome 28
Time Frame: 0 to 30 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

64. Secondary Outcome: Freedom From Ipsilateral Major Amputation
Description: as for outcome 28
Time Frame: 0 to 180 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

65. Secondary Outcome: Freedom From Ipsilateral Major Amputation
Description: as for outcome 28
Time Frame: 0 to 365 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

66. Secondary Outcome: Freedom From Ipsilateral Major Amputation
Description: as for outcome 28
Time Frame: 0 to 379 days
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 141
percentage of participants | 100

67. Secondary Outcome: Quality of Life Measures : Physical Functioning (PF)
Description: SF-12 Norm-Based Scores; Quality of Life (SF-12®) is a standardized, validated questionnaire used to evaluate general health outcomes. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible.
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 115
score on a scale | 41.53 (11.83)

68. Secondary Outcome: Quality of Life Measures : Physical Functioning (PF)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 41.70 (12.06)

69. Secondary Outcome: Quality of Life Measures : Physical Functioning (PF)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 38.28 (11.85)

70. Secondary Outcome: Quality of Life Measures : Role Physical (RP)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 116
score on a scale | 43.83 (10.26)

71. Secondary Outcome: Quality of Life Measures : Role Physical (RP)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 42.94 (11.86)

72. Secondary Outcome: Quality of Life Measures : Role Physical (RP)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 109
score on a scale | 41.07 (11.50)

73. Secondary Outcome: Quality of Life Measures : Bodily Pain (BP)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 116
score on a scale | 43.83 (12.09)

74. Secondary Outcome: Quality of Life Measures : Bodily Pain (BP)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 41.52 (13.15)

75. Secondary Outcome: Quality of Life Measures : Bodily Pain (BP)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 109
score on a scale | 42.30 (12.06)

76. Secondary Outcome: Quality of Life Measures : General Health (GH)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 117
score on a scale | 38.49 (9.24)

77. Secondary Outcome: Quality of Life Measures : General Health (GH)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 39.72 (10.20)

78. Secondary Outcome: Quality of Life Measures : General Health (GH)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 39.65 (9.50)

79. Secondary Outcome: Quality of Life Measures : Vitality (VT)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 117
score on a scale | 46.89 (11.49)

80. Secondary Outcome: Quality of Life Measures : Vitality (VT)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 47.83 (11.14)

81. Secondary Outcome: Quality of Life Measures : Vitality (VT)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 46.57 (11.49)

82. Secondary Outcome: Quality of Life Measures : Social Functioning (SF)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 117
score on a scale | 49.40 (9.84)

83. Secondary Outcome: Quality of Life Measures : Social Functioning (SF)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 47.47 (12.80)

84. Secondary Outcome: Quality of Life Measures : Social Functioning (SF)
Description: SF-12 Norm-Based Scores; Quality of Life (SF-12®) is a standardized, validated questionnaire used to evaluate general health outcomes. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible.
  rm-Based Scores.
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 48.74 (10.69)

85. Secondary Outcome: Quality of Life Measures : Role Emotional (RE)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 117
score on a scale | 46.86 (11.94)

86. Secondary Outcome: Quality of Life Measures : Role Emotional (RE)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 119
score on a scale | 45.79 (12.22)

87. Secondary Outcome: Quality of Life Measures : Role Emotional (RE)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 109
score on a scale | 45.97 (12.11)

88. Secondary Outcome: Quality of Life Measures : Mental Health (MH)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 117
score on a scale | 50.94 (10.42)

89. Secondary Outcome: Quality of Life Measures : Mental Health (MH)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 121
score on a scale | 50.44 (10.79)

90. Secondary Outcome: Quality of Life Measures : Mental Health (MH)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 50.10 (11.18)

91. Secondary Outcome: Quality of Life Measures : Physical Component Summary (PCS)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 114
score on a scale | 39.82 (9.99)

92. Secondary Outcome: Quality of Life Measures : Physical Component Summary (PCS)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 119
score on a scale | 39.71 (11.11)

93. Secondary Outcome: Quality of Life Measures : Physical Component Summary (PCS)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 109
score on a scale | 37.51 (10.75)

94. Secondary Outcome: Quality of Life Measures : Mental Component Summary (MCS)
Description: as for outcome 67
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 114
score on a scale | 52.03 (9.99)

95. Secondary Outcome: Quality of Life Measures : Mental Component Summary (MCS)
Description: as for outcome 67
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 119
score on a scale | 51.08 (10.36)

96. Secondary Outcome: Quality of Life Measures : Mental Component Summary (MCS)
Description: as for outcome 67
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 109
score on a scale | 51.71 (10.38)

97. Secondary Outcome: Vascular Quality of Life (VascuQol) Total Scores
Description: Vascular Quality of Life (VascuQol) : A standardized, validated questionnaire used to evaluate vascular disease-specific health outcomes. VascuQol total score includes scores of Activity Domain, Symptom Domain, Pain Domain, Emotional Domain and Social Domain. Each item is rated as a 7 point response scale, with a score of 1 being the worst and a score of 7 the best possible. The total average score is the sum of all 25 items scores divided by 25. For each separate domain an average score can be calculated (sum of all items of one domain divided by the number of items of that domain). The highest score for each domain is 7, which indicates best health outcome.
  There are no sub scales.
Time Frame: 1 month
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 120
score on a scale | 5.62 (1.37)

98. Secondary Outcome: Vascular Quality of Life (VascuQol) Total Scores
Description: as for outcome 97
Time Frame: 6 months
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 124
score on a scale | 5.38 (1.55)

99. Secondary Outcome: Vascular Quality of Life (VascuQol) Total Scores
Description: as for outcome 97
Time Frame: 1 year
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Number analyzed (Participants) | 111
score on a scale | 5.41 (1.36)

ADVERSE EVENTS:
Time Frame: 12 months (365 days)
Arm/Group | Absolute Pro® and Pro LL® Peripheral Stent Systems
Serious Adverse Events (participants affected / at risk) | 81/141
Other Adverse Events (participants affected / at risk) | 95/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absolute Pro® and Pro LL® Peripheral Stent Systems (N=141)
Hematoma (Injury, poisoning and procedural complications) | 1
Allergic Reaction To Diabetic Meds (Immune system disorders) | 1
other (Immune system disorders) | 2
Rash (Immune system disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 2
Abnormal Lab Test (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Pancreatic Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angina (Cardiac disorders) | 4
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 8
CAD - Coronary stenosis (Cardiac disorders) | 2
Cardiac Arrest (Cardiac disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 4
Hypertension (Cardiac disorders) | 1
Myocardial Infarction - Non Q wave (Cardiac disorders) | 2
Myocardial Infarction - Unknown (Cardiac disorders) | 1
Myocardial Infarction ST Elevated (Cardiac disorders) | 1
Other (Cardiac disorders) | 10
Pain (Cardiac disorders) | 10
Surgery/Intervention Procedure (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
(Cardiac disorders) | 1
Ventricular Dysfunction (Cardiac disorders) | 1
Cholecystitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
GI Bleed (Gastrointestinal disorders) | 1
Other (Gastrointestinal disorders) | 2
Pain (Gastrointestinal disorders) | 1
Kidney Damage Due To Other (Renal and urinary disorders) | 1
Pyelonephritis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Urinary Tract Infection (Renal and urinary disorders) | 1
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pancreatic Disorder (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 1
Wound Complication Or Wound Infection (Infections and infestations) | 2
Encephalopathy (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Other (Metabolism and nutrition disorders) | 1
Abnormal Lab Test (Investigations) | 1
Other (Investigations) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Other (Musculoskeletal and connective tissue disorders) | 1
Surgery/Intervention Procedure (Musculoskeletal and connective tissue disorders) | 2
Trauma (Musculoskeletal and connective tissue disorders) | 1
Depression (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Ischemic Encephalopathy (Nervous system disorders) | 1
Mental Status Change (Nervous system disorders) | 4
Other (Nervous system disorders) | 1
Edema (Non Pulmonary) (Surgical and medical procedures) | 1
Pseudoaneurysm (Surgical and medical procedures) | 1
Asbestosis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 3
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Lung Mass (Respiratory, thoracic and mediastinal disorders) | 1
Malignant (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Ischemic Stroke (Nervous system disorders) | 1
(Nervous system disorders) | 4
Claudication (Vascular disorders) | 8
Embolism (Vascular disorders) | 1
Hematoma (Vascular disorders) | 2
Ischemia (Vascular disorders) | 1
Occlusion (Vascular disorders) | 1
PAD (Vascular disorders) | 1
PVD (Vascular disorders) | 9
Pseudoaneurysm (Vascular disorders) | 3
Pulmonary Emboli (Vascular disorders) | 1
Pulmonary Embolism (Vascular disorders) | 1
Renal Artery Disease (Vascular disorders) | 1
Restenosis (Vascular disorders) | 19
Stenosis (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Absolute Pro® and Pro LL® Peripheral Stent Systems (N=141)
Arrhythmia (Includes Brady And Tachy) (Cardiac disorders) | 12
Pain (General disorders) | 13
Pain (Musculoskeletal and connective tissue disorders) | 15
Claudication (Vascular disorders) | 17
Peripheral vascular diseases (PVD) (Vascular disorders) | 17
Restenosis (Vascular disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days